CLINICAL TRIAL: NCT02887274
Title: Application of Stimulated Immune Response Change to Predict Outcome of Patient With Severe Sepsis
Acronym: SIRCSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG8B1073
Record Dates: First submitted 2016-08-15; First posted 2016-09-02 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-08

CONDITIONS: Systemic Inflammatory Response Syndrome (SIRS); Sepsis; Severe Sepsis; Septic Shock; Multiple Organ Failure
Keywords: Systemic Inflammatory Response Syndrome (SIRS); Sepsis; Severe Sepsis; Septic shock; Multiple organ failure
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum immunological biomarkers including cytokines, blood cell counts, and biochemistry profiles.
Oversight: Data Monitoring Committee: No

SUMMARY:
Persistence of a marked compensatory anti-inflammatory innate immune response after an insult is termed immunoparalysis. There is no biomarker available to determine the immune status of patient. Thus, the need for early and definite diagnosis of immune status of patient with sepsis, as well as the identification of patients at risk of evolving with severe organ dysfunctions, is crucial.

Most important of all, speed is the key to survival. Therefore, it of crucial importance to identify which patient characteristic determines the poor prognosis. Early intervention can improve the prognosis. Investigators foresee an urgent need to identify predictors for mortality in severe sepsis, including clinical factors or immune status. Recently, the PIRO model has been proposed as a way of stratifying septic patients according to their Predisposing condition, the severity of Infection, the Response to therapy and the degree of Organ dysfunction. The immune status may be associated with above model. However, there is paucity data addressing this issue. In this study, investigators will also analyze the progression of patient condition during treatment and the associated immune status change. In the future, Investigators hope the determination of immune status may contribute to this model of classification rather than just being used as prognostic markers. Despite the advances in the knowledge of the basic processes that trigger and sustain the systemic inflammatory response in sepsis, the search for a "magic bullet" to treat this syndrome has been frustrating. The incidence of severe sepsis and septic shock still remains quite high, as does its mortality, which has decreased very little over the past decades.

DETAILED DESCRIPTION:
Binding of TLRs to epitopes on microorganisms stimulates intracellular signaling, increasing transcription of proinflammatory molecules such as tumor necrosis factor α (TNF-α) and interleukin-1β, as well as antiinflammatory cytokines such as interleukin-10. Macrophage dysfunction, as a component of immune suppression seen during trauma and sepsis, appears to be one of the contributing factors to morbidity and mortality. Critically ill patients demonstrating prolonged, severe reductions in monocyte HLA-DR expression or ex vivo tumor necrosis factor alpha production are at high risk for nosocomial infection and death. Most septic patients have decreasing cytokine levels at the time of treatment, suggesting a transition from a hyperinflammatory to a hypo-inflammatory state. Immunoparalysis is a potentially reversible risk factor for development of nosocomial infection in multiple organ dysfunction syndrome. Whole-blood ex vivo TNF alpha response is a promising marker for monitoring this condition. Investigators call it as "stimulated immune response". Toll-like receptors (TLRs) are a recently described family of immune receptors involved in the recognition of pathogen-associated molecular patterns (PAMPs). Lipopolysaccharide (LPS) is present in the outer membranes of Gram-negative bacteria and has been demonstrated to be responsible for the development of GNB-associated sepsis. Recognition of bacterial LPS by macrophages is a key component of host defense against infection by Gram-negative bacteria. A monocyte which encounters LPS should vigorously produce proinflammatory cytokines regardless of whether or not it has been exposed to LPS in the past. Sepsis induces suppression of macrophage function as determined by a reduction of pro-inflammatory cytokine production upon re-exposure to lipopolysaccharide (LPS) in vitro. Whether further ground can be gained by manipulating innate immunity is an important question waiting to be answered. Several strategies to enhance innate immunity have been tried in normal subjects, including using granulocyte colony-stimulating factor to increase the number and activation state of circulating neutrophils, and IFN-γ to enhance macrophage dependent immunity. Investigators will use this characteristic to assess patient's stimulated immune response. In addition, differences in the nature of the initiating agent causing sepsis and the lack of co-morbidities in the animal models probably contribute to some of the differences in animal studies and clinical trials in sepsis. Investigators need to address these important issues and work toward promoting immunologic homeostasis in the ICU. Here investigators performed a systematic study aimed at evaluating

1. The diagnostic accuracy of stimulated immune response for predicting mortality;
2. Whether trend change in stimulated immune response more useful for above prediction;
3. Whether stimulated immune response can predict patients at risk of evolving with severe organ dysfunctions (the presence or development of severe sepsis or progression of organ dysfunctions within a 72-hr time period from biomarker checked along with treatment)

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis
* Septic shock

Exclusion Criteria:

* Patients are < 18 yrs
* Patients are immunocompromised (treatment with corticosteroids >1 mg/kg equivalent prednisone)
* Bone marrow or organ transplant recipients,
* Leucopenia [white blood cells count< 109/L] or neutropenia [polymorphonuclear granulocyte count <0.5 109/L]
* Hematologic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at Kaohsiung Chang Gung Memorial Hospital. All adult patients presenting with sepsis or severe sepsis will be enrolled on admission to medical intensive units (total 34 beds). Sepsis and severe sepsis are defined as American College of Chest Physicians/Society of Critical Care Medicine consensus criteria for sepsis syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of stimulated immune response for predicting mortality | 4 weeks, up to 24 weeks

SECONDARY OUTCOMES:
Whether trend change in stimulated immune response more useful for prediction mortality | 4 weeks, up to 24 weeks

OTHER OUTCOMES:
Whether stimulated immune response can predict patients at risk of evolving with severe organ dysfunctions | 4 weeks, up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Feng Fang, M.D, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Frazier WJ, Hall MW. Immunoparalysis and adverse outcomes from critical illness. Pediatr Clin North Am. 2008 Jun;55(3):647-68, xi. doi: 10.1016/j.pcl.2008.02.009. PMID 18501759
- [Result] Hall MW, Knatz NL, Vetterly C, Tomarello S, Wewers MD, Volk HD, Carcillo JA. Immunoparalysis and nosocomial infection in children with multiple organ dysfunction syndrome. Intensive Care Med. 2011 Mar;37(3):525-32. doi: 10.1007/s00134-010-2088-x. Epub 2010 Dec 10. PMID 21153402
- [Result] Neveu H, Kleinknecht D, Brivet F, Loirat P, Landais P. Prognostic factors in acute renal failure due to sepsis. Results of a prospective multicentre study. The French Study Group on Acute Renal Failure. Nephrol Dial Transplant. 1996 Feb;11(2):293-9. doi: 10.1093/oxfordjournals.ndt.a027256. PMID 8700363
- [Result] Vincent JL, Abraham E, Annane D, Bernard G, Rivers E, Van den Berghe G. Reducing mortality in sepsis: new directions. Crit Care. 2002 Dec;6 Suppl 3(Suppl 3):S1-18. doi: 10.1186/cc1860. Epub 2002 Dec 5. PMID 12720570
- [Result] Marshall JC, Charbonney E, Gonzalez PD. The immune system in critical illness. Clin Chest Med. 2008 Dec;29(4):605-16, vii. doi: 10.1016/j.ccm.2008.08.001. PMID 18954696
- [Result] Sakr Y, Burgett U, Nacul FE, Reinhart K, Brunkhorst F. Lipopolysaccharide binding protein in a surgical intensive care unit: a marker of sepsis? Crit Care Med. 2008 Jul;36(7):2014-22. doi: 10.1097/CCM.0b013e31817b86e3. PMID 18552695
- [Result] Shiramizo SC, Marra AR, Durao MS, Paes AT, Edmond MB, Pavao dos Santos OF. Decreasing mortality in severe sepsis and septic shock patients by implementing a sepsis bundle in a hospital setting. PLoS One. 2011;6(11):e26790. doi: 10.1371/journal.pone.0026790. Epub 2011 Nov 3. PMID 22073193
- [Result] Nguyen HB, Corbett SW, Steele R, Banta J, Clark RT, Hayes SR, Edwards J, Cho TW, Wittlake WA. Implementation of a bundle of quality indicators for the early management of severe sepsis and septic shock is associated with decreased mortality. Crit Care Med. 2007 Apr;35(4):1105-12. doi: 10.1097/01.CCM.0000259463.33848.3D. PMID 17334251
- [Result] Phua J, Koh Y, Du B, Tang YQ, Divatia JV, Tan CC, Gomersall CD, Faruq MO, Shrestha BR, Gia Binh N, Arabi YM, Salahuddin N, Wahyuprajitno B, Tu ML, Wahab AY, Hameed AA, Nishimura M, Procyshyn M, Chan YH; MOSAICS Study Group. Management of severe sepsis in patients admitted to Asian intensive care units: prospective cohort study. BMJ. 2011 Jun 13;342:d3245. doi: 10.1136/bmj.d3245. PMID 21669950
- [Result] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500